CLINICAL TRIAL: NCT06040216
Title: Long-term Follow-up Results of Ectopic Inner Foveal Retinal Layers Evolution Following Pars Plana Vitrectomy
Brief Title: Evolution of EIFL Following PPV
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Levent Karabas, Prof. Dr., Kocaeli University
Other Study IDs: KocaeliUniversity
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stage 2 ERM
  Interventions: Other: optical coherence tomography
- Stage 3 ERM
  Interventions: Other: optical coherence tomography
- Stage 4 ERM
  Interventions: Other: optical coherence tomography

INTERVENTIONS:
Other: optical coherence tomography — We observed the postoperative improvement in EIFL severity with optical coherence tomography

SUMMARY:
Various classification systems have been described for epiretinal membrane (ERM). One of them is a new OCT-based staging scheme based on displacement and reorganization of inner retinal layers called ectopic inner retinal layers (EIFL). We evaluated pre-and perioperative factors related to time for evolution of EIFL.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing idiopathic epiretinal membrane surgery

Exclusion Criteria:

* Patients undergoing seconder epiretinal membrane surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study included 81 consecutive eyes with idiopathic epiretinal membrane that underwent vitrectomy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 1-month
  Best corrected visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University School of Medicine, Kocaeli, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No